CLINICAL TRIAL: NCT02244515
Title: Consequence of Dexmedetomidine on Emergence Deliruim After Sevoflurane Anesthesia in Children With Cerebral Palsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jin Ni (Other)
Responsible Party: Sponsor-Investigator, Jin Ni, Vice-administrator of Department of Anesthesiology, Guangzhou Women and Children's Medical Center
Organization: Guangzhou Women and Children's Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ED cerebral palsy
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Emergence Deliruim; Cerebral Palsy
Keywords: children
MeSH Terms: conditions — Cerebral Palsy | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Group C (Placebo Comparator): Five minutes prior to the commencement of the surgical procedure, Group D participants were administered 10 ml NaCI 0.9%.
- Group D (Experimental): Five minutes prior to the commencement of the surgical procedure, Group D participants were administered dexmedetomidine 0.5μg•kg-1 diluted in 10 ml NaCI 0.9%
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine 0.5μg•kg-1 diluted in 10 ml NaCI 0.9%
  Arms: Group D

SUMMARY:
The purpose of this study is to determine whether dexmedetomidine is effective in the treatment of emergence deliruim after sevoflurane anesthesia in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

Non-quadriplegic (mono-,di-, hemiplegic) children with CP that are scheduled for elective Achilles-tendon lengthening procedure Guangzhou Women and Children's Medical Center, Guangzhou, China, with American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

Participants that displayed symptoms of sinus bradycardia and atrio-ventricular block, non-communicative severe developmental delay, seizure disorders, and treatment with seizure medications

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
pediatric anesthesia emergence delirium (PAED) scale | during stay in postanesthesia care unit
Heart rate | during surgical procedures
systolic blood pressure | during surgical procedures
diastolic blood pressure | during surgical procedures